CLINICAL TRIAL: NCT05346796
Title: Survivorship Plan HEalth REcord (SPHERE) Implementation Trial
Acronym: SPHERE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David A. Haggstrom, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10523; 1R01CA241143-01A1 (NIH)
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Group that will receive written survivorship care information.
- Intervention (Experimental): Group that will be provided access to the survivorship care plan-personal health record tool.
  Interventions: Behavioral: Survivorship Care Plan-Personal Health Record (SCP-PHR)

INTERVENTIONS:
Behavioral: Survivorship Care Plan-Personal Health Record (SCP-PHR) — The SCP-PHR tool is an online portal that is intended to help cancer survivors manage their survivorship care.
  Arms: Intervention

SUMMARY:
To understand the effectiveness and implementation of the SCP-PHR, we will conduct a hybrid type 1 effectiveness-implementation trial consisting of the following components: (A) a randomized clinical effectiveness trial, and (B) a mixed methods implementation study.

DETAILED DESCRIPTION:
The Institute of Medicine recommends that each cancer patient receive a survivorship care plan that summarizes information important to the individual's long-term care, including the following: (1) cancer type and treatments, (2) their potential consequences, (3) recommendations regarding preventive practices, and (4) specific information about recommended follow-up. Despite their clinical importance, gaps in colorectal cancer (CRC) surveillance care and preventive care exist among CRC survivors. Unmet symptom needs are also prevalent and undertreated.

We propose to evaluate the capacity of an interactive survivorship care plan (SCP) delivered through an Internet-based personal health record (PHR) to meet the needs of CRC survivors. PHRs combine health information and medical data with knowledge management and software tools to potentially enable patients to become active participants in their own care. A SCP delivered via an appropriately designed PHR may promote increased concordance with CRC surveillance and preventive care guidelines through the exchange of health information with CRC survivors. A survivorship care plan-personal health record (SCP-PHR) may also improve care for symptoms through the combination of longitudinal PHR- based symptom measurement and tailored self-management tools. To understand the effectiveness of the SCP-PHR, we will conduct a randomized clinical effectiveness trial at the patient level. We will assess impact of the SCP-PHR across a variety of measures and outcomes, including CRC surveillance, preventive care receipt, patient symptoms, and patient-centered quality.

To simultaneously understand the effectiveness and implementation of the SCP-PHR, we will conduct a hybrid type I effectiveness-implementation trial consisting of the following components: (A) a randomized clinical effectiveness trial at the patient level, and (B) a mixed methods implementation study. The mixed methods portion of the study will consist of a qualitative process evaluation using semi- structured interviews to assess facilitators and barriers to implementation of the SCP-PHR among key stakeholders: patients, health care providers, and organizational leaders. This study design will enable us to meet the simultaneous needs of understanding the effectiveness and the health care context of SCP implementation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years or older at the time of consent
2. Patients must have regular (at least weekly) access to an internet connection, whether at home or elsewhere (family or friend).
3. Diagnosis of colon or rectal cancer, Stages I, II, or III (AJCC, American Joint Committee on Cancer) and have undergone initial curative-intent therapy for their CRC diagnosis within the past 12 months.
4. English-speaking

Exclusion Criteria:

1. Patient will be excluded if they have had recurrence of their colorectal cancer.
2. Patient's with severe cognitive impairment
3. Patient's with schizophrenia or other psychosis
4. Patients currently in hospice care

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Colorectal Cancer Surveillance Outcomes | 12 months
  The CRC Surveillance Index (SI) will be extracted from the electronic medical record. For each observation period, every person-month is classified as either "covered" (eligible for the test during the month and covered) or "uncovered" (eligible for the test, but not covered). If a surveillance test (S) is delivered to an eligible patient at a particular time, then all person-months for the following recommended interval fall under a period of coverage (P1). If it is not renewed, then an uncovered portion of the observation period (U) is created. Further, if a second surveillance test (S2) is performed after some uncovered interval (U), additional covered months (P2) may be present during the observation period. For each patient, SI=100*[(P1+P2)/(P1+P2+U)] for each surveillance test.

SECONDARY OUTCOMES:
Preventive Care Outcomes | 12 months
  All preventive care measures will be measured in the electronic medical record based upon U.S. Preventive Services Task Force (USPSTF) or Advisory Committee for Immunization Practices guidelines. Measures are calculated using a methodology similar to the one described for the Surveillance Index, but in this instance, a Prevention Index (PI) is created. The following preventive care is included in the index: influenza vaccine, pneumococcal vaccine, cholesterol screening, blood pressure screening, and HIV screening screening118, tobacco status and counseling119, screening mammography119, and cervical cancer screening
Symptom Measures | 12 months
  The primary symptom outcome measure will be the composite 5-symptom T score from the PROMIS which includes scales for sleep, pain, anxiety, depression, and energy/fatigue (SPADE) via self-report. Conversion tables allow conversion of simple summed raw scores from PROMIS scales into T-score values. The composite Patient-Reported Outcomes Measurement Information System (PROMIS) score is the mean of the 5 symptom scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States